CLINICAL TRIAL: NCT03673670
Title: A Phase II, Randomized, Double Blind, Placebo Controlled, Three-way Crossover Study to Assess the Bronchodilator Effect of RPL554 Administered in Addition to Open Label Tiotropium/Olodaterol in Patients With COPD
Brief Title: Bronchodilator Effect of RPL554 Administered in Addition to Tiotropium/Olodaterol in Patients With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RPL554-CO-204
Record Dates: First submitted 2018-09-07; First posted 2018-09-17 (Actual); Results first posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-09

CONDITIONS: COPD
Keywords: COPD; Bronchodilation; FEV1
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The nebulizer cup will be obscured so the contents are not visible to the subject and the blinded study staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1.5 mg RPL554 and tiotropium/olodaterol (Experimental): 1.5 mg RPL554 suspension administered using a nebulizer twice daily plus 5 mcg/5 mcg tiotropium/olodaterol (Respimat) administered once daily
  Interventions: Drug: RPL554 Suspension; Drug: Tiotropium/olodaterol (Respimat)
- 6 mg RPL554 and tiotropium/olodaterol (Experimental): 6 mg RPL554 suspension administered using a nebulizer twice daily plus 5 mcg/5 mcg tiotropium/olodaterol (Respimat) administered once daily
  Interventions: Drug: RPL554 Suspension; Drug: Tiotropium/olodaterol (Respimat)
- Placebo and tiotropium/olodaterol (Experimental): Placebo administered using a nebulizer twice daily plus 5 mcg/5 mcg tiotropium/olodaterol (Respimat) administered once daily
  Interventions: Drug: Placebo; Drug: Tiotropium/olodaterol (Respimat)

INTERVENTIONS:
Drug: RPL554 Suspension — A PDE3/4 inhibitor
  Arms: 1.5 mg RPL554 and tiotropium/olodaterol; 6 mg RPL554 and tiotropium/olodaterol
Drug: Placebo — A placebo solution
  Arms: Placebo and tiotropium/olodaterol
Drug: Tiotropium/olodaterol (Respimat) — An anticholinergic/β-agonist combination medication

SUMMARY:
The study investigates the effect of 3 days of twice daily treatment of two different doses of RPL554 (a phosphodiesterase [PDE]3/4 inhibitor) or placebo, each administered in addition to once daily tiotropium/olodaterol (Respimat) in patients with moderate to severe chronic obstructive pulmonary disease (COPD). Patients will receive each of the three treatment combinations in a randomized sequence using a crossover design

DETAILED DESCRIPTION:
RPL554 is a dual inhibitor of phosphodiesterase 3 (PDE3) and phosphodiesterase 4 (PDE4) which are known to have a role in modulating the inflammatory airway response in respiratory diseases, including COPD. PDE3 inhibitors act as bronchodilators whilst PDE4 inhibitors have anti-inflammatory properties and there is also evidence to suggest that combined inhibition of PDE3 and PDE4 can have additive or synergistic anti-inflammatory and bronchodilator. The two doses of RPL554 (1.5 mg and 6 mg)have been selected based on the results from prior studies investigating single and multiple ascending doses in healthy subjects, single doses in asthmatics, single/multiple ascending doses in COPD patients, and 3 days of dosing in COPD patients. These doses were demonstrated to be both effective as a bronchodilator and well tolerated.

The purpose of the study is to investigate if RPL554 has an additive bronchodilator effect when administered in combination with a commonly used anticholinergic/β-agonist combination medication, tiotropium/olodaterol (Respimat), in this patient population measured by the peak forced expiratory volume in one second (FEV1), and forced vital capacity (FVC).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Male or female aged 40 and 80 years
3. For males, not to donate sperm and either be sexually abstinent or use contraception as specified by the protocol. For females, be of non-childbearing potential or use a highly effective form of contraception
4. 12-lead ECG with heart rate between 45 and 90 beats per minute, QTcF ≤450 msec for males, and ≤ 470 msec for females, QRS interval ≤120 msec and no clinically significant abnormality including morphology
5. Screening Holter report with a minimum of 18 hours recording that is able to be evaluated for rhythm analysis showing no abnormality which indicates a significant impairment of patient safety or which may significantly impair interpretation
6. Capable of complying with all study restrictions and procedures including ability to use the study nebulizer and Respimat® correctly.
7. Body mass index (BMI) between 18 and 36 kg/m2 and minimum weight of 45 kg.
8. COPD diagnosis for at least 1 year and clinically stable COPD for 4 week
9. Post-bronchodilator (two puffs of salbutamol/albuterol followed by two puffs of ipratropium) spirometry at Screening:

   * Post-bronchodilator FEV1/forced vital capacity (FVC) ratio of ≤0.70
   * Post-bronchodilator FEV1 ≥30 % and ≤70% of predicted normal
   * Demonstrates ≥150 mL increase from pre-bronchodilator FEV1
10. A chest X-ray showing no abnormalities, which are both clinically significant and unrelated to COPD.

12. Meet the concomitant medication restrictions and be expected to do so for the rest of the study.

13. Current and former smokers with smoking history of ≥10 pack years. 14. Capable of withdrawing from long acting bronchodilators for the duration of the study, and short acting bronchodilators for 8 hours prior to dosing.

Exclusion Criteria:

1. A history of life-threatening COPD including Intensive Care Unit admission and/or requiring intubation.
2. COPD exacerbation requiring oral or parenteral steroids, or lower respiratory tract infection requiring antibiotics, in the last 3 months
3. A history of one or more hospitalizations for COPD in the last 12 months
4. Intolerance or hypersensitivity to tiotropium, olodaterol, atropine, ipratropium, or RPL554.
5. Evidence of cor pulmonale or clinically significant pulmonary hypertension.
6. Other respiratory disorders
7. Previous lung resection or lung reduction surgery.
8. Use of oral COPD medications, except mucolytics, in the last 3 months
9. Pulmonary rehabilitation, unless such treatment has been stable in the last 4 weeks
10. History of, or reason to believe a patient has, drug or alcohol abuse within the past 5 years.
11. Inability to perform acceptable spirometry or whole body plethysmography
12. Received an experimental drug within 30 days or five half lives, whichever is longer.
13. Patients with uncontrolled disease that the Investigator believes are clinically significant. This includes any hepatic disease, or an alanine aminotransferase or aspartate aminotransferase>2 x upper limit of normal (ULN).
14. Documented cardiovascular disease: arrhythmias, angina, recent (<1 year) or suspected myocardial infarction, congestive heart failure, unstable or uncontrolled hypertension, or diagnosis of hypertension in the last 3 months
15. Use of non-selective oral β-blockers.
16. Major surgery (requiring general anesthesia) in the last 6 weeks or will not have fully recovered from surgery, or planned surgery through the end of the study.
17. A disclosed history or one known to the Investigator, of significant non compliance in previous investigational studies or with prescribed medications.
18. Required use of oxygen therapy, even on an occasional basis.
19. Symptomatic prostatic hyperplasia or bladder-neck obstruction or with narrow-angle glaucoma.
20. History of malignancy of any organ system within 5 years, with the exception of localized skin cancers (basal or squamous cell).
21. Clinically significant abnormal values for safety laboratory tests (hematology, biochemistry, virology or urinalysis) as determined by the Investigator
22. Any other reason that the Investigator considers makes the patient unsuitable to participate.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, Principal Investigator — Medicines Evaluation Unit
Locations (4):
- United States (2):
  - Clinical Site Partners, LLC, Winter Park, Florida
  - Allied Biomedical Research Holdings, d/b/a Vitalink Research, Greenville, South Carolina
- United Kingdom (2):
  - Respiratory Clinical Trials LTD,, London
  - Medicines Evaluation Unit, Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose RPL554 Then High Dose RPL554 Then Placebo: 1.5 mg RPL554 twice daily plus tiotropium 5/5 mcg once daily for 3 days then 6 mg RPL554 twice daily plus tiotropium 5/5 mcg once daily for 3 days then placebo twice daily plus tiotropium 5/5 mcg once daily for 3 days with a 7-14 day washout between treatment periods
- Low Dose RPL554 Then Placebo Then High Dose RPL554: 1.5 mg RPL554 twice daily plus tiotropium 5/5 mcg once daily for 3 days then placebo twice daily plus tiotropium 5/5 mcg once daily for 3 days then 6 mg RPL554 twice daily plus tiotropium 5/5 mcg once daily for 3 days with a 7-14 day washout between treatment periods
- High Dose RPL554 Then Low Dose RPL554 Then Placebo: 6 mg RPL554 twice daily plus tiotropium 5/5 mcg once daily for 3 days then 1.5 mg RPL554 twice daily plus tiotropium 5/5 mcg once daily for 3 days then placebo twice daily plus tiotropium 5/5 mcg once daily for 3 days with a 7-14 day washout between treatment periods
- High Dose RPL554 Then Placebo Then Low Dose RPL554: 6 mg RPL554 twice daily plus tiotropium 5/5 mcg once daily for 3 days then placebo twice daily plus tiotropium 5/5 mcg once daily for 3 days then 1.5 mg RPL554 twice daily plus tiotropium 5/5 mcg once daily for 3 days with a 7-14 day washout between treatment periods
- Placebo Then Low Dose RPL554 Then High Dose RPL554: Placebo twice daily plus tiotropium 5/5 mcg once daily for 3 days then 1.5 mg RPL554 twice daily plus tiotropium 5/5 mcg once daily for 3 days then 6 mg RPL554 twice daily plus tiotropium 5/5 mcg once daily for 3 days with a 7-14 day washout between treatment periods
- Placebo Then High Dose RPL554 Then Low Dose RPL554: Placebo twice daily plus tiotropium 5/5 mcg once daily for 3 days then 6 mg RPL554 twice daily plus tiotropium 5/5 mcg once daily for 3 days then 1.5 mg RPL554 twice daily plus tiotropium 5/5 mcg once daily for 3 days with a 7-14 day washout between treatment periods
Period: Treatment Period 1 (3 Days)
Arm/Group | Low Dose RPL554 Then High Dose RPL554 Then Placebo | Low Dose RPL554 Then Placebo Then High Dose RPL554 | High Dose RPL554 Then Low Dose RPL554 Then Placebo | High Dose RPL554 Then Placebo Then Low Dose RPL554 | Placebo Then Low Dose RPL554 Then High Dose RPL554 | Placebo Then High Dose RPL554 Then Low Dose RPL554
Started | 14 | 14 | 13 | 12 | 13 | 13
Completed | 13 | 14 | 12 | 12 | 13 | 11
Not Completed | 1 | 0 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Alpha 1 antitrypsin deficiency | 0 | 0 | 0 | 0 | 0 | 1
Period: Washout Period 1 (7-14 Days)
Arm/Group | Low Dose RPL554 Then High Dose RPL554 Then Placebo | Low Dose RPL554 Then Placebo Then High Dose RPL554 | High Dose RPL554 Then Low Dose RPL554 Then Placebo | High Dose RPL554 Then Placebo Then Low Dose RPL554 | Placebo Then Low Dose RPL554 Then High Dose RPL554 | Placebo Then High Dose RPL554 Then Low Dose RPL554
Started | 13 | 14 | 12 | 12 | 13 | 11
Completed | 13 | 14 | 12 | 12 | 13 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (3 Days)
Arm/Group | Low Dose RPL554 Then High Dose RPL554 Then Placebo | Low Dose RPL554 Then Placebo Then High Dose RPL554 | High Dose RPL554 Then Low Dose RPL554 Then Placebo | High Dose RPL554 Then Placebo Then Low Dose RPL554 | Placebo Then Low Dose RPL554 Then High Dose RPL554 | Placebo Then High Dose RPL554 Then Low Dose RPL554
Started | 13 | 14 | 12 | 12 | 13 | 11
Completed | 13 | 14 | 11 | 12 | 12 | 11
Not Completed | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 0
Period: Washout Period 2 (7-14 Days)
Arm/Group | Low Dose RPL554 Then High Dose RPL554 Then Placebo | Low Dose RPL554 Then Placebo Then High Dose RPL554 | High Dose RPL554 Then Low Dose RPL554 Then Placebo | High Dose RPL554 Then Placebo Then Low Dose RPL554 | Placebo Then Low Dose RPL554 Then High Dose RPL554 | Placebo Then High Dose RPL554 Then Low Dose RPL554
Started | 13 | 14 | 11 | 12 | 12 | 11
Completed | 13 | 14 | 11 | 12 | 11 | 11
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Pre-dose FEV1 not 20% baseline | 0 | 0 | 0 | 0 | 1 | 0
Period: Treatment Period 3 (3 Days)
Arm/Group | Low Dose RPL554 Then High Dose RPL554 Then Placebo | Low Dose RPL554 Then Placebo Then High Dose RPL554 | High Dose RPL554 Then Low Dose RPL554 Then Placebo | High Dose RPL554 Then Placebo Then Low Dose RPL554 | Placebo Then Low Dose RPL554 Then High Dose RPL554 | Placebo Then High Dose RPL554 Then Low Dose RPL554
Started | 13 | 14 | 11 | 12 | 11 | 11
Completed | 13 | 14 | 11 | 12 | 10 | 11
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose RPL554 Then High Dose RPL554 Then Placebo | Low Dose RPL554 Then Placebo Then High Dose RPL554 | High Dose RPL554 Then Low Dose RPL554 Then Placebo | High Dose RPL554 Then Placebo Then Low Dose RPL554 | Placebo Then Low Dose RPL554 Then High Dose RPL554 | Placebo Then High Dose RPL554 Then Low Dose RPL554 | Total
Number analyzed (Participants) | 14 | 14 | 13 | 12 | 13 | 13 | 79
Age, Continuous [Median (Full Range); unit: years] | 65.5 [43 to 75] | 64.5 [53 to 74] | 63.0 [45 to 74] | 63.0 [43 to 77] | 67.0 [49 to 76] | 61.0 [48 to 73] | 64.0 [43 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 8 | 7 | 8 | 8 | 49
  Male | 5 | 5 | 5 | 5 | 5 | 5 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 1 | 1 | 2 | 0 | 1 | 6
  White | 13 | 13 | 12 | 10 | 13 | 11 | 72
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peak FEV1 on Day 3
Description: Change from baseline FEV1 to peak FEV1 (measured as the greatest value in the 4 hours post-dose after the morning dose) on Day 3
Time Frame: Change from pre-dose at 5, 15 and 30 minutes and 1, 1.5, 2 & 4 hours on Day 3
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 1.5 mg RPL554 and Tiotropium/Olodaterol | 6 mg RPL554 and Tiotropium/Olodaterol | Placebo and Tiotropium/Olodaterol
Number analyzed (Participants) | 74 | 73 | 73
Liters | 0.565 (0.2783) | 0.506 (0.2506) | 0.519 (0.2809)
Statistical Analysis 1: Comparison: 1.5 mg RPL554 and Tiotropium/Olodaterol vs Placebo and Tiotropium/Olodaterol; Test type: Other — A hierarchical fixed-sequence testing strategy was employed to test the significance of the treatment effect for each of the two RPL554 doses against placebo, starting with the highest dose (6 mg). If a statistically significant difference was found at the 2-sided α level of 5%, the testing proceeded with the next highest dose. Otherwise, testing was stopped, and the remaining null hypotheses were accepted without testing; p = 0.168, ANCOVA; GeoMean Ratio = 1.021, 95% CI 2-sided [0.991 to 1.052]
Statistical Analysis 2: Comparison: 6 mg RPL554 and Tiotropium/Olodaterol vs Placebo and Tiotropium/Olodaterol; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.731, ANCOVA; GeoMean Ratio = 0.995, 95% CI 2-sided [0.966 to 1.025]

2. Secondary Outcome: Change From Baseline to Trough FEV1 on Day 4
Description: Change from baseline to morning trough FEV1 on Day 4
Time Frame: Change from pre-dose on Day 1 to pre-dose on Day 4
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 1.5 mg RPL554 and Tiotropium/Olodaterol | 6 mg RPL554 and Tiotropium/Olodaterol | Placebo and Tiotropium/Olodaterol
Number analyzed (Participants) | 74 | 73 | 73
Liters | 0.186 (0.2496) | 0.178 (0.2123) | 0.150 (0.2218)
Statistical Analysis 1: Comparison: 1.5 mg RPL554 and Tiotropium/Olodaterol vs Placebo and Tiotropium/Olodaterol; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.115, ANCOVA; GeoMean Ratio = 1.024, 95% CI 2-sided [0.994 to 1.055]
Statistical Analysis 2: Comparison: 6 mg RPL554 and Tiotropium/Olodaterol vs Placebo and Tiotropium/Olodaterol; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.111, ANCOVA; GeoMean Ratio = 1.024, 95% CI 2-sided [0.994 to 1.055]

3. Secondary Outcome: Change From Baseline in AUC0-4h FEV1 on Day 3
Description: Change from baseline FEV1 to AUC FEV1 over 4 hours post-dose after the morning dose on Day 3. The endpoint is measured as AUC/interval length (average) and measured in liters. (Note: Endpoint is AUC/interval length (average) so the units are in liters.)
Time Frame: Change from pre-dose to each of the following timepoints: 5, 15 and 30 minutes and 1, 1.5, 2, 4 hours on Day 3 (after the morning dose)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 1.5 mg RPL554 and Tiotropium/Olodaterol | 6 mg RPL554 and Tiotropium/Olodaterol | Placebo and Tiotropium/Olodaterol
Number analyzed (Participants) | 74 | 73 | 73
Liters | 0.429 (0.2518) | 0.390 (0.2246) | 0.377 (0.2485)
Statistical Analysis 1: Comparison: 6 mg RPL554 and Tiotropium/Olodaterol vs Placebo and Tiotropium/Olodaterol; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.303, ANCOVA; GeoMean Ratio = 1.014, 95% CI 2-sided [0.987 to 1.043]

4. Secondary Outcome: Change From Baseline in AUC0-12h FEV1 on Day 3
Description: Change from baseline in AUC over 12 hours post-dose after the morning dose on Day 3. The endpoint is measured as AUC/interval length (average) and measured in liters (Note: Endpoint is AUC/interval length (average) so the units are in liters.)
Time Frame: Change from pre-dose to each of the following timepoints: 5, 15 and 30 minutes and 1, 1.5, 2, 4, 6, 8, 12 hours on Day 3 (after the morning dose)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 1.5 mg RPL554 and Tiotropium/Olodaterol | 6 mg RPL554 and Tiotropium/Olodaterol | Placebo and Tiotropium/Olodaterol
Number analyzed (Participants) | 74 | 73 | 73
Liters | 0.390 (0.2426) | 0.347 (0.2219) | 0.337 (0.2447)
Statistical Analysis 1: Comparison: 1.5 mg RPL554 and Tiotropium/Olodaterol vs Placebo and Tiotropium/Olodaterol; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.067, ANCOVA; GeoMean Ratio = 1.027, 95% CI 2-sided [0.998 to 1.057]
Statistical Analysis 2: Comparison: 6 mg RPL554 and Tiotropium/Olodaterol vs Placebo and Tiotropium/Olodaterol; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.395, ANCOVA; GeoMean Ratio = 1.012, 95% CI 2-sided [0.984 to 1.042]

5. Secondary Outcome: Change From Baseline in Peak FEV1 on Day 1
Description: Change from baseline FEV1 to peak FEV1 in the 4 hours post-dose after the morning dose on Day 1
Time Frame: Change from pre-dose to each of the following timepoints: 5, 15 and 30 minutes and 1, 1.5, 2, 4 hours on Day 1 (after the morning dose), with the maximum change reported
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 1.5 mg RPL554 and Tiotropium/Olodaterol | 6 mg RPL554 and Tiotropium/Olodaterol | Placebo and Tiotropium/Olodaterol
Number analyzed (Participants) | 74 | 73 | 73
Liters | 0.490 (0.2219) | 0.467 (0.2393) | 0.445 (0.2306)
Statistical Analysis 1: Comparison: 6 mg RPL554 and Tiotropium/Olodaterol vs Placebo and Tiotropium/Olodaterol; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.404, ANCOVA; GeoMean Ratio = 1.012, 95% CI 2-sided [0.984 to 1.039]

6. Secondary Outcome: Change From Baseline in Peak FEV1 After Evening Dose on Day 3
Description: Change from baseline FEV1 to peak FEV1 in the 4 hours post-dose after the evening dose on Day 3
Time Frame: Change from pre-dose to each of the ollowing timepoints: 5, 15 and 30 minutes and 1, 1.5, 2, 4 hours on Day 3 (after the evening dose), with the maximum change reported
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 1.5 mg RPL554 and Tiotropium/Olodaterol | 6 mg RPL554 and Tiotropium/Olodaterol | Placebo and Tiotropium/Olodaterol
Number analyzed (Participants) | 74 | 73 | 73
Liters | 0.453 (0.2625) | 0.405 (0.2581) | 0.324 (0.2211)
Statistical Analysis 1: Comparison: 1.5 mg RPL554 and Tiotropium/Olodaterol vs Placebo and Tiotropium/Olodaterol; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.001, ANCOVA; GeoMean Ratio = 1.082, 95% CI 2-sided [1.043 to 1.123]
Statistical Analysis 2: Comparison: 6 mg RPL554 and Tiotropium/Olodaterol vs Placebo and Tiotropium/Olodaterol; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.002, ANCOVA; GeoMean Ratio = 1.061, 95% CI 2-sided [1.023 to 1.101]

7. Secondary Outcome: Change From Baseline in AUC0-12h FEV1 on Day 1
Description: Change from baseline FEV1 to AUC FEV1 over 12 hours post-dose after the morning dose on Day 1. The endpoint is measured as AUC/interval length (average) and measured in liters (Note: Endpoint is AUC/interval length (average) so the units are in liters.)
Time Frame: Change from pre-dose to each of the following timepoints: 5, 15 and 30 minutes and 1, 1.5, 2, 4, 6, 8, 12 hours on Day 1 (after the morning dose)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 1.5 mg RPL554 and Tiotropium/Olodaterol | 6 mg RPL554 and Tiotropium/Olodaterol | Placebo and Tiotropium/Olodaterol
Number analyzed (Participants) | 74 | 73 | 73
Liters | 0.333 (0.1815) | 0.308 (0.1854) | 0.303 (0.1920)
Statistical Analysis 1: Comparison: 1.5 mg RPL554 and Tiotropium/Olodaterol vs Placebo and Tiotropium/Olodaterol; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.096, ANCOVA; GeoMean Ratio = 1.020, 95% CI 2-sided [0.997 to 1.043]
Statistical Analysis 2: Comparison: 6 mg RPL554 and Tiotropium/Olodaterol vs Placebo and Tiotropium/Olodaterol; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.862, ANCOVA; GeoMean Ratio = 1.002, 95% CI 2-sided [0.979 to 1.025]

8. Secondary Outcome: Determination of Onset of Action on Day 1
Description: Time to >10% increase in FEV1 from pre-first dose, censored at 2 hours
Time Frame: Change from pre-dose to the following timepoints: 5, 15 and 30 minutes and 1, 1.5, 2 hours on Day 1 (after the morning dose)
Population: Full analysis set
Measure: Median (Full Range); unit: minutes
Arm/Group | 1.5 mg RPL554 and Tiotropium/Olodaterol | 6 mg RPL554 and Tiotropium/Olodaterol | Placebo and Tiotropium/Olodaterol
Number analyzed (Participants) | 74 | 73 | 73
minutes | 10.0 [1 to 86] | 6.0 [4 to 117] | 11.0 [7 to 120]
Statistical Analysis 1: Comparison: 1.5 mg RPL554 and Tiotropium/Olodaterol vs Placebo and Tiotropium/Olodaterol; Test type: Other; p = 0.945, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0
Statistical Analysis 2: Comparison: 6 mg RPL554 and Tiotropium/Olodaterol vs Placebo and Tiotropium/Olodaterol; Test type: Other; p = 0.501, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0

9. Secondary Outcome: Residual Volume on Day 1
Description: Change in residual volume during treatment
Time Frame: Change from pre-dose to 1.25 hours on Day 1 (after the morning dose)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- 1.5 mg RPL554 and Tiotropium/Olodaterol on Day 1: 1.5 mg RPL554 suspension administered using a nebulizer twice daily plus 5 mcg/5 mcg tiotropium/olodaterol (Respimat) administered once daily
  RPL554 Suspension: A PDE3/4 inhibitor
  Tiotropium/olodaterol (Respimat): An anticholinergic/β-agonist combination medication
- 6 mg RPL554 and Tiotropium/Olodaterol on Day 1: 6 mg RPL554 suspension administered using a nebulizer twice daily plus 5 mcg/5 mcg tiotropium/olodaterol (Respimat) administered once daily
  RPL554 Suspension: A PDE3/4 inhibitor
  Tiotropium/olodaterol (Respimat): An anticholinergic/β-agonist combination medication
- Placebo and Tiotropium/Olodaterol on Day 1: Placebo administered using a nebulizer twice daily plus 5 mcg/5 mcg tiotropium/olodaterol (Respimat) administered once daily
  Placebo: A placebo solution
  Tiotropium/olodaterol (Respimat): An anticholinergic/β-agonist combination medication
Arm/Group | 1.5 mg RPL554 and Tiotropium/Olodaterol on Day 1 | 6 mg RPL554 and Tiotropium/Olodaterol on Day 1 | Placebo and Tiotropium/Olodaterol on Day 1
Number analyzed (Participants) | 74 | 73 | 74
Liters | -0.469 (0.5521) | -0.408 (0.4803) | -0.377 (0.4810)

10. Secondary Outcome: Residual Volume on Day 3
Description: Change in residual volume during treatment
Time Frame: Change from pre-dose on Day 1 to the following timepoints: pre-dose, 1.25, 8.25 and 12.25 hours on Day 3 (after the morning dose)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- 1.5 mg RPL554 and Tiotropium/Olodaterol on Day 3: 1.5 mg RPL554 suspension administered using a nebulizer twice daily plus 5 mcg/5 mcg tiotropium/olodaterol (Respimat) administered once daily
  RPL554 Suspension: A PDE3/4 inhibitor
  Tiotropium/olodaterol (Respimat): An anticholinergic/β-agonist combination medication
- 6 mg RPL554 and Tiotropium/Olodaterol on Day 3: 6 mg RPL554 suspension administered using a nebulizer twice daily plus 5 mcg/5 mcg tiotropium/olodaterol (Respimat) administered once daily
  RPL554 Suspension: A PDE3/4 inhibitor
  Tiotropium/olodaterol (Respimat): An anticholinergic/β-agonist combination medication
- Placebo and Tiotropium/Olodaterol on Day 3: Placebo administered using a nebulizer twice daily plus 5 mcg/5 mcg tiotropium/olodaterol (Respimat) administered once daily
  Placebo: A placebo solution
  Tiotropium/olodaterol (Respimat): An anticholinergic/β-agonist combination medication
Arm/Group | 1.5 mg RPL554 and Tiotropium/Olodaterol on Day 3 | 6 mg RPL554 and Tiotropium/Olodaterol on Day 3 | Placebo and Tiotropium/Olodaterol on Day 3
Number analyzed (Participants) | 74 | 73 | 73
Liters
  Pre-dose Day 3 | -0.323 (0.4548) | -0.313 (0.8946) | -0.184 (0.6274)
  1.25 hours | -0.648 (0.5173) | -0.510 (0.6304) | -0.510 (0.6257)
  8.25 hours | -0.526 (0.5594) | -0.481 (0.4994) | -0.471 (0.6186)
  12.25 hours | -0.353 (0.4561) | -0.236 (0.7566) | -0.094 (0.7118)

11. Secondary Outcome: Functional Residual Capacity on Day 1
Description: Change in functional residual capacity during treatment
Time Frame: Change from pre-dose to 1.25 hours on Day 1 (after the morning dose)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 1.5 mg RPL554 and Tiotropium/Olodaterol on Day 1 | 6 mg RPL554 and Tiotropium/Olodaterol on Day 1 | Placebo and Tiotropium/Olodaterol on Day 1
Number analyzed (Participants) | 74 | 73 | 73
Liters | -0.344 (0.5097) | -0.294 (0.4524) | -0.277 (0.4279)

12. Secondary Outcome: Functional Residual Capacity on Day 3
Description: Change in functional residual capacity during treatment
Time Frame: as for outcome 10
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- 1.5 mg RPL554 and Tiotropium/Oldaterol on Day 3: 1.5 mg RPL554 suspension administered using a nebulizer twice daily plus 5 mcg/5 mcg tiotropium/olodaterol (Respimat) administered once daily
  RPL554 Suspension: A PDE3/4 inhibitor
  Tiotropium/olodaterol (Respimat): An anticholinergic/β-agonist combination medication
- 6 mg RPL554 and Tiotropium/Oldaterol on Day 3: 6 mg RPL554 suspension administered using a nebulizer twice daily plus 5 mcg/5 mcg tiotropium/olodaterol (Respimat) administered once daily
  RPL554 Suspension: A PDE3/4 inhibitor
  Tiotropium/olodaterol (Respimat): An anticholinergic/β-agonist combination medication
- Placebo and Tiotropium/Oldaterol on Day 3: Placebo administered using a nebulizer twice daily plus 5 mcg/5 mcg tiotropium/olodaterol (Respimat) administered once daily
  Placebo: A placebo solution
  Tiotropium/olodaterol (Respimat): An anticholinergic/β-agonist combination medication
Arm/Group | 1.5 mg RPL554 and Tiotropium/Oldaterol on Day 3 | 6 mg RPL554 and Tiotropium/Oldaterol on Day 3 | Placebo and Tiotropium/Oldaterol on Day 3
Number analyzed (Participants) | 74 | 73 | 73
Liters
  1.25 hours | -0.490 (0.4654) | -0.408 (0.6102) | -0.382 (0.5610)
  8.25 hours | -0.420 (0.5003) | -0.405 (0.6111) | -0.355 (0.6004)
  12.25 hours | -0.255 (0.4003) | -0.155 (0.7788) | -0.075 (0.5881)
  Pre-dose on Day 3 | -0.278 (0.4340) | -0.206 (0.5925) | -0.163 (0.5742)

13. Secondary Outcome: Specific Airway Conductance on Day 1
Description: Change in specific airway conductance during treatment
Time Frame: Change from pre-dose to 1.25 hours on Day 1 (after the morning dose)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: 1/kPa*sec
Arm/Group | 1.5 mg RPL554 and Tiotropium/Olodaterol on Day 1 | 6 mg RPL554 and Tiotropium/Olodaterol on Day 1 | Placebo and Tiotropium/Olodaterol on Day 1
Number analyzed (Participants) | 74 | 73 | 73
1/kPa*sec | 0.064 (0.1148) | 0.042 (0.0483) | 0.043 (0.1072)

14. Secondary Outcome: Specific Airway Conductance on Day 3
Description: Change in specific airway conductance during treatment
Time Frame: as for outcome 10
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: 1/kPa*sec
Arm/Group | 1.5 mg RPL554 and Tiotropium/Olodaterol on Day 3 | 6 mg RPL554 and Tiotropium/Olodaterol on Day 3 | Placebo and Tiotropium/Olodaterol on Day 3
Number analyzed (Participants) | 74 | 73 | 73
1/kPa*sec
  Pre-dose Day 3 | 0.021 (0.608) | 0.046 (0.1060) | 0.016 (0.0890)
  1.25 hours | 0.064 (0.0824) | 0.050 (0.0682) | 0.049 (0.1193)
  8.25 hours | 0.059 (0.1312) | 0.048 (0.0733) | 0.037 (0.1125)
  12.25 hours | 0.029 (0.0774) | 0.032 (0.0629) | 0.021 (0.1071)

ADVERSE EVENTS:
Time Frame: From informed consent until the end of the study, approximately 2 months for each patient
Description: As this is a cross over study, the number of patients at risk for each event was specified as the total number of patients who received the specified treatment in either Treatment Period 1, 2 or 3.
Arm/Group | 1.5 mg RPL554 and Tiotropium/Olodaterol | 6 mg RPL554 and Tiotropium/Olodaterol | Placebo and Tiotropium/Olodaterol
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/74 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/75 | 1/74 | 0/76
Other Adverse Events (participants affected / at risk) | 15/75 | 15/74 | 8/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.5 mg RPL554 and Tiotropium/Olodaterol (N=75) | 6 mg RPL554 and Tiotropium/Olodaterol (N=74) | Placebo and Tiotropium/Olodaterol (N=76)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1.5 mg RPL554 and Tiotropium/Olodaterol (N=75) | 6 mg RPL554 and Tiotropium/Olodaterol (N=74) | Placebo and Tiotropium/Olodaterol (N=76)
Headache (Nervous system disorders) | 5 | 5 | 1
Ventricular extrasystoles (Cardiac disorders) | 2 | 3 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Hypertension (Vascular disorders) | 0 | 2 | 1
syncope (Nervous system disorders) | 0 | 0 | 1
Accelerated idioventricular rhythm (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 0
Medical device site rash (General disorders) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall not be permitted to present at symposia, national or regional professional meetings, and to publish in journals, theses or dissertations, or otherwise of their own choosing, methods and results of the Clinical Trial subject to the publication policy described in the Protocol without prior written approval of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-05-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT03673670/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT03673670/SAP_001.pdf